Official Title: The effects of spasticity on glucose metabolism and soft tissue body

composition in individuals with motor complete and motor incomplete spinal cord

injury

NCT03859960

Document date: August 6th, 2020

## **INFORMED CONSENT FORM**

In our study "The relationship between spasticity and glucose metabolism in patients with spinal cord injury", it is aimed to investigate whether there is a relationship between spasticity and blood sugar levels. Patients who accept to participate in the study will be examined, their spasticity will be evaluated, and height, weight, hip and waist circumference will be measured. Body fat ratio and lean mass ratios will be measured with the Bone Densitometry device. After taking fasting blood, 75 grams of glucose should be diluted and patients will drink it for sugar loading test. The patients' blood samples in the quantity of 2 ml will be taken before the loading glucose and then 30, 60, 90, and 120 minutes after taking the glucose solution to measure the serum glucose and insulin levels. Blood will be drawn again at 30, 60, 90 and 120 minutes after glucose is ingested. Nausea and temporary vomiting may occur during the sugar loading test. The amount of radiation to be taken with Bone Densitometry is very low. If you agree to participate in the study, there is no other risk. You will not be charged any fees for all examinations, tests and other medical care covered by this study. If any abnormality is found in the laboratory tests, your treatment will be started early. Also, the results drawn from this study can be used for the benefit of other people. If you do not agree to participate in this study, you are entitled to accepted treatments.

## **VOLUNTEER APPROVAL FORM**

The above information about this research was given to me by stating that a medical research will be conducted in Fatih Sultan Mehmet Training and Research Hospital Physical Medicine and Rehabilitation Department by Dr. Arzu Atici. After this information, I was invited as a "participant" (subject) to such a study. If I participate in this research, I believe that the confidentiality of my information that should remain between me and the physician will be approached with great care and respect during this research. I have been given sufficient confidence that my personal information will be protected with care when using research results for educational and scientific purposes. I can withdraw from the research without

giving any reason during the execution of the project. I can also be excluded from research by the researcher, provided that my medical condition is not harmed. I do not take any financial responsibility for the expenses for research. No payment will be made to me either. I understand all the explanations given to me in detail. I made the decision to take part in this research project as a "participant" (subject). I accept the invitation on this subject with great satisfaction and willingness. A copy of this signed form sheet will be given to me. Name-Surname, Signature, Address of the Volunteer (telephone number, fax number, if any) Name-surname, Signature, Address of the parent or guardian for those under guardianship or guardianship (telephone number, fax number, if any) Name-surname, Signature of the researcher who made the explanations. Name, Surname, Signature, Duty of the organization officer who witnessed the process from the beginning to the end.